CLINICAL TRIAL: NCT04539379
Title: Evaluation of Intravenous Infusion of Labetalol Versus Magnesium Sulfate on Cerebral Hemodynamics of Severe Preeclampsia Patients Using Transcranial Doppler
Brief Title: Evaluation of Intravenous Infusion of Labetalol Versus Magnesium Sulfate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, lecture of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6353
Record Dates: First submitted 2020-08-30; First posted 2020-09-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Magnesium Sulfate; Labetalol
Keywords: magnesium sulfate, labetalol, severe preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate; Labetalol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium sulfate (Active Comparator): intravenous infusion of magnesium sulfate at a dose of 4 gm intravenously over 20 min as a loading dose then MgSO4 intravenous infusion is continued at a rate of 1 gm/h for 24 h or until obtain and stabilize the targeted blood pressure..
  Interventions: Drug: Magnesium sulfate
- labetolol (Active Comparator): The patients will be given intravenous infusion of labetolol (Trandate™, 5mg/ml) available in 20 ml ampoules containing 100mg labetalol (5mg/ml). Starting the infusion with 20mg/h and then titrate to obtain and stabilize the targeted blood pressure by adjusting the infusion as required every 15 - 30min to a maximum dose of 160mg/hr.
  Interventions: Drug: Labetolol

INTERVENTIONS:
Drug: Magnesium sulfate — intravenous infusion
  Arms: magnesium sulfate
Drug: Labetolol — intravenous infusion
  Other Names: (Trandate™,)
  Arms: labetolol

SUMMARY:
the purpose of this study is to compare Intravenous infusion of Labetalol versus Magnesium Sulfate on Cerebral Hemodynamics of Severe Preeclampsia Patients using Transcranial Doppler

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double blind manner into 2 groups each one containing 30 patients , (Group M) : will be given intravenous infusion of magnesium sulfate at a dose of 4 gm intravenously over 20 min as a loading dose then MgSO4 intravenous infusion is continued at a rate of 1 gm/h for 24 h or until obtain and stabilize the targeted blood pressure..

(Group L) : The patients will be given intravenous infusion of labetalol (Trandate™,) available in 20 ml ampoules containing 100mg labetalol (5mg/ml). Starting the infusion with 20mg/h and then titrate to obtain and stabilize the targeted blood pressure by adjusting the infusion as required every 15 - 30min to a maximum dose of 160mg/hr.

ELIGIBILITY:
Inclusion Criteria:

* acceptance
* 21 to 45 years old.
* mass index ≤ 35 kg/m2.
* Singleton Pregnant female complicated with severe preeclampsia
* Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 110 mmHg on two occasions at least 4 hours apart
* Thrombocytopenia (platelet count less than 100,000 )
* Impaired liver function indicated by elevated liver enzymes (to twice the upper limit normal concentration), and severe persistent right upper quadrant or epigastric pain not responding to medications and not explained by another diagnosis.
* Renal insufficiency (serum creatinine concentration more than 1.1 mg/dL or doubling of the serum creatinine concentration in the absence of other renal disease)
* Pulmonary edema
* New-onset headache unresponsive to medications and not accounted for by alternative diagnoses
* Visual disturbances.

Exclusion Criteria:

* Preexisting heart disease
* Known pulmonary disorders.
* Inadequate temporal window.
* Atrial fibrillation and any rhythm abnormality.
* History of allergy or contraindications to either magnesium sulfate or labetolol.
* Exposure to any of the study medications within 24 hours of enrollment.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Singleton Pregnant female complicated with severe preeclampsia
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
mean velocity | basal measurements before administration of the study drugs then at post-treatment one and six hours after drug administration.
  mean velocity of middle cerebral artery

SECONDARY OUTCOMES:
mean end diastolic velocity | basal measurements before administration of the study drugs then at post-treatment one and six hours after drug administration.
  mean end diastolic velocity of middle cerebral artery
pulsatility index | basal measurements before administration of the study drugs then at post-treatment one and six hours after drug administration.
  pulsatility index of middle cerebral artery
cerebral perfusion pressure | basal measurements before administration of the study drugs then at post-treatment one and six hours after drug administration.
  cerebral perfusion pressure
occurrence of seizures | basal measurements before administration of the study drugs then at post-treatment one and six hours after drug administration.
  occurrence of seizures
The need for other antihypertensive drugs | post-treatment one and six hours after drug administration.
  The need for other antihypertensive drugs (nifidibine, nitroglycerine, hydralazine, etc)
adverse effects of the study drugs | post-treatment till 24 hours
  hypotension,Bradycardia,persistent hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Howida A kamal, M.D, Study Director — zagazig U
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Zagazig, Elsharkia,egypt, Egypt

REFERENCES:
- [Derived] Mowafy SMS, Medhat MM. Evaluation of intravenous infusion of labetalol versus magnesium sulfate on cerebral hemodynamics of preeclampsia patients with severe features using transcranial doppler. J Clin Monit Comput. 2023 Aug;37(4):951-961. doi: 10.1007/s10877-023-01006-4. Epub 2023 Apr 19. PMID 37074522